CLINICAL TRIAL: NCT03080220
Title: Effects of Pre-Event Soft Tissue Treatment on Functional Movement and Functional Performance
Brief Title: Examining the Effects of Three Soft Tissue Treatments on Functional Movement and Functional Performance Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rocky Mountain University of Health Professions (Other)
Collaborators: Performance Dynamics (Unknown); Indiana Athletic Trainers' Association (Unknown)
Responsible Party: Principal Investigator, Andrew Doyle, Associate Professor at Indiana Wesleyan University, Rocky Mountain University of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 160231-03
Record Dates: First submitted 2017-03-11; First posted 2017-03-15 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Functional Performance
MeSH Terms: interventions — Canes; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Astym (Experimental): The Astym treatment (AT) is specifically used by medical professionals to treat musculoskeletal dysfunctions by stimulating the body's ability to break down adhesions and reabsorb dysfunctional tissue (scar tissue).6-16,19 The treatment induces collagen building, fibroblastic activity, and phagocytosis.17,18 Part of the treatment includes utilizing a series of instruments glided across the skin tissue, in a non-invasive manner, along the route of the underlying muscle fibers' direction. The treatment specifically spares healthy tissue and stimulates growth factors and cellular mediators that stimulate the repair of dysfunctional tissue in the body's internal mechanisms.17,18 Astym is an FDA approved device. Specifically, Astym is registered as having a device class as 1 and regulation number as 890.5660.
  Interventions: Device: Astym
- Stick (Experimental): The Stick treatment (ST) utilizes an instrument to convert non-compliant muscle to compliant muscle by compressing the muscle. The individual spindles of The Stick create a stripping massage by applying progressively deeper strokes over the soft tissue.38 The Stick permits individuals to perform trigger point release on own person, allowing the muscle to become compliant to the wanted movement.
  Interventions: Device: Stick
- Massage (Placebo Comparator): Similar to the protocol previously outlined for the other two independent variables, the massage treatment (MT) will progress from anterior, to medial, to lateral and posterior shank, thigh, and hip. The treatment on each muscle tissue will follow the similar protocol as the Astym treatment (AT) group. However, the flat, non-treatment edge of the Evaluator®, Localizer®, and Isolator® will be put in contact with the muscle tissues in a direction parallel to the muscle fibers being treated, but without over pressure.7 The traditional treatment edge of the instrument has a tapered, machine edge and creates shear forces when glided across the tissue at an angle between 60 and 80 degrees.
  Interventions: Device: Massage

INTERVENTIONS:
Device: Astym — therapeutic massage instrument
  Arms: Astym
Device: Stick — massage instrument
  Other Names: The Stick
  Arms: Stick
Device: Massage — massage instruments
  Arms: Massage

SUMMARY:
The purpose of this study is to investigate the effects of Astym® treatment, The Stick® treatment and massage treatment on performance among healthy college athletes and to investigate any relationship between functional movement and functional performance. Participants will be recruited from Division II, National Association of Intercollegiate Athletics (NAIA) basketball and volleyball teams. The participants will be randomized into one of three groups: Astym treatment (AT), The Stick treatment (ST) or massage treatment (MT). The participant will have baseline measures of vertical jump (VJ), Y-Balance Lower Quarter Screen (YBLQ), and a rating of current perceived lower extremity function using a visual analog scale (PLEF-VAS). The participants will be treated using either the AT, ST, or MT following baseline measures. Immediately following the intervention, a second measurement of VJ, YBLQ, and PLEF-VAS will take place. The data will be analyzed using mixed ANOVA tests which will be conducted for each dependent variable. In addition, functional movement is thought to be related to functional performance. A Pearson Product Correlation analysis will be used to understand any relationship between YBLQ and VJ. It is hypothesized that those in the AT group will have different percent change in their YBLQ, VJ, and PLEF-VAS compared to those in ST and MT groups. It is hypothesized that a correlation between YBLQ and VJ will exist. As a result, clinicians could use AT among basketball and volleyball athletes without hindering acute performance. Any risks the participants could encounter are minimal. Participants may withdraw themselves and their data at any time. The intervention and testing are similar to what an athlete would be exposed to during their collegiate career. Any participant injured during this study will be referred to their university sports medicine staff, health center, or the Indiana Wesleyan University health center.

DETAILED DESCRIPTION:
All participants will complete baseline testing, intervention, and post intervention testing in a single day. The total time for a participant to complete the entire study is anticipated to be between 1.5 and 2 hours. Upon arrival to the Athletic Training Clinic, a participant's demographic information will be collected. This information will consist of the following: age, weight, height, and percent body fat using a standard seven site skinfold measurement. Other information will be recorded, such as sport, position, gender, years of college sport experience, and year in school. The research team will ensure that the participant is dressed appropriately in athletic shorts and T-shirt. Spandex® or compression type garments will not be allowed to be worn at any time during the study.

Once the demographic information is collected, a full body warm up will be initiated. Participants will be instructed to warm up on a bike for 5 minutes at an intensity of 4 to 6 as represented on the OMNI scale of perceived exertion. This warm up is based on the guidelines set forth by the American College of Sports Medicine. Following the warm up, each participant's baseline measurements will be taken in this order: Vertical Jump (VJ), Y-Balance Lower Quarter (YBLQ), and rating of Perceived Lower Extremity Function-Visual Analog Scale (PLEF-VAS).

Following baseline data collection, participants will be randomly assigned to an intervention. One of the three treatments previously described will take place in the Athletic Training Clinic. An individual not associated with the research committee or research team will conduct the randomization. Immediately following the intervention, participants will proceed to the performance evaluation testing area for post treatment testing. The participant may elect to bring one chaperon of their choosing to the treatment area. Warm up and performance testing order will remain consistent for each participant and will follow the order as conducted during baseline measure.

Trained undergraduate research assistants, blinded from the treatment allocation will collect the testing data. The testing data will include: the VJ, YBLQ, and the PLEF-VAS. The clinicians (doctoral candidate and assisting clinician) will provide Astym treatment (AT), The Stick treatment (ST), or massage treatment (MT) and will not be present for the VJ, YBLQ, and the PLEF-VAS nor will the clinicians providing the intervention be present in the testing area during baseline test collection.

Testing Procedures Participants will perform the VJ and YBLQ Screen following a 5-minute-warm up as previously described. The highest jump of three attempts will be recorded for the counter movement VJ. The longest reach of three attempts in the anterior, posteriolateral and posteromedial directions will be recorded following the established YBLQ protocol.

Vertical Jump A Belt Mat (University of Toronto; Toronto, Canada) vertical jump measuring device will be utilized for this study. The participant is positioned on a mat with a belt placed around the waist. The belt has a tape measure running form the belt to the mat. The participant is asked to stand erect to establish 'zero'. The participant then jumps vertically while the belt is around the waist pulling out the remaining tape measure. The vertical jump height is recorded as the displacement of the tape measure. The participant will propel vertically as high as possible. A preparatory stutter step will not be used; however, a counter movement may be used. A countermovement is where the participant quickly flexes the knees and hips while moving the thorax forward and downward while swinging the arms back. Three jump attempts will be given to each participant where a measurement will take place after each attempt. Measurements will be recorded to the nearest half inch and then converted to centimeters. The highest measurement will be used for analysis.

Y Balance Lower Quarter Screen Testing procedures for the YBLQ (Y Balance Test Kit, Move2Perform; Evansville, IN) will follow the protocol previously established by researchers The participant will have viewed a two minute instructional video prior to practicing six reaches in each of the three directions bilaterally: anterior, posteriormedial and posteriorlateral. Following the practice reaches, the participant will stand on the Y Balance center footplate with the right foot behind the start line. With the free foot, the participant will reach in the anterior direction pushing the indicator box as far as possible. Three successful measurements in as many as six attempts in the reach direction will be recorded with the best, successful reach being used for analysis. The participant will then switch stance legs. The indicator box will be reset and the participant will reach with the right foot in the anterior direction. This cycle will continue for the posteromedial and posterolateral directions. Successful reaches are those where the participant maintained contact with stance leg on the center footplate and behind the start line throughout the reach attempt. Successful reaches also will include maintaining contact with the indicator box during the reach attempt, not using the indicator box for support, and returning to start position under control. The participant will rest only as long as it takes the recorder to reset the indicator box and log the reach distance.

Rating of Perceived Lower Extremity Function The participant will be asked to rate current perceived lower extremity function on a 100mm line anywhere between 'my function is at its worst' and 'my function is at its best.' The participant will rate by placing a vertical line that intersects the 100mm horizontal line perpendicularly. A standard metric ruler will be used to measure from the farthest left to the intersecting line. This distance will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* male and female athletes
* individuals aged between 18 and 25 years
* compete in basketball or volleyball sponsored by the NAIA Division II governing body during the 2015 - 2016 or 2016 - 2017 athletic seasons
* sport eligible.

Exclusion Criteria:

* Astym treatment (AT) in last 3 weeks
* The Stick treatment (ST) in the last 3 weeks
* Massage treatment (MT) in thelast 3 weeks
* Participants using other means of instrument assisted cutaneous tissue preparation techniques such as 'scraping' household items or stainless steel objects along the lower kinetic chain tissue.
* Currently injured or ill
* Injured in the last month before the participation date
* Not full healed from a previous injury or illness
* Participants who currently have athletic participation restrictions of any kind - Those who have known clotting dysfunctions
* Those on anticoagulation therapies
* Those with neurogenic dysfunctions
* Those who may be pregnant
* Those allergic to cocoa butter.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | 1 day
  A Belt Mat (University of Toronto; Toronto, Canada) vertical jump measuring device will be utilized for this study.28
Dynamic Balance | 1 day
  A Y Balance test kit will be used to measure the distance reached while the participant stabilizes on one leg.

SECONDARY OUTCOMES:
Rating of Perceived Lower Extremity Function | 1 day
  The participant will be asked to rate current perceived lower extremity function on a 100mm line anywhere between 'my function is at its worst' and 'my function is at its best.' The participant will rate by placing a vertical line that intersects the 100mm horizontal line perpendicularly. A standard metric ruler will be used to measure from the farthest left to the intersecting line. This distance will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Doyle, MA, Principal Investigator — Rocky Mountain University of Health Professions/Indiana Wesleyan University
Locations (3):
- United States (3):
  - University of Saint Francis, Fort Wayne, Indiana
  - Huntington University, Huntington, Indiana
  - Indiana Wesleyan University, Marion, Indiana

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this point.

REFERENCES:
- [Background] Mikesky AE, Bahamonde RE, Stanton K, Alvey T, Fitton T. Acute effects of The Stick on strength, power, and flexibility. J Strength Cond Res. 2002 Aug;16(3):446-50. PMID 12173961
- [Background] Healey KC, Hatfield DL, Blanpied P, Dorfman LR, Riebe D. The effects of myofascial release with foam rolling on performance. J Strength Cond Res. 2014 Jan;28(1):61-8. doi: 10.1519/JSC.0b013e3182956569. PMID 23588488
- [Background] Fletcher IM. The effects of precompetition massage on the kinematic parameters of 20-m sprint performance. J Strength Cond Res. 2010 May;24(5):1179-83. doi: 10.1519/JSC.0b013e3181ceec0f. PMID 20386129
- [Background] Goodwin JE, Glaister M, Howatson G, Lockey RA, McInnes G. Effect of pre-performance lower-limb massage on thirty-meter sprint running. J Strength Cond Res. 2007 Nov;21(4):1028-31. doi: 10.1519/R-20275.1. PMID 18076229
- [Background] Arroyo-Morales M, Fernandez-Lao C, Ariza-Garcia A, Toro-Velasco C, Winters M, Diaz-Rodriguez L, Cantarero-Villanueva I, Huijbregts P, Fernandez-De-las-Penas C. Psychophysiological effects of preperformance massage before isokinetic exercise. J Strength Cond Res. 2011 Feb;25(2):481-8. doi: 10.1519/JSC.0b013e3181e83a47. PMID 21240029
- [Background] Sevier TL, Stegink-Jansen CW. Astym treatment vs. eccentric exercise for lateral elbow tendinopathy: a randomized controlled clinical trial. PeerJ. 2015 May 19;3:e967. doi: 10.7717/peerj.967. eCollection 2015. PMID 26038722
- [Background] Kivlan BR, Carcia CR, Clemente FR, Phelps AL, Martin RL. The effect of Astym(R) Therapy on muscle strength: a blinded, randomized, clinically controlled trial. BMC Musculoskelet Disord. 2015 Oct 29;16:325. doi: 10.1186/s12891-015-0778-9. PMID 26510526
- [Background] Chughtai M, Mont MA, Cherian C, Cherian JJ, Elmallah RD, Naziri Q, Harwin SF, Bhave A. A Novel, Nonoperative Treatment Demonstrates Success for Stiff Total Knee Arthroplasty after Failure of Conventional Therapy. J Knee Surg. 2016 Apr;29(3):188-93. doi: 10.1055/s-0035-1569482. Epub 2015 Dec 29. PMID 26713596
- [Background] Slaven EJ, Mathers J. Management of chronic ankle pain using joint mobilization and ASTYM(R) treatment: a case report. J Man Manip Ther. 2011 May;19(2):108-12. doi: 10.1179/2042618611Y.0000000004. PMID 22547921
- [Background] McCormack JR. The management of bilateral high hamstring tendinopathy with ASTYM(R) treatment and eccentric exercise: a case report. J Man Manip Ther. 2012 Aug;20(3):142-6. doi: 10.1179/2042618612Y.0000000003. PMID 23904753
- [Background] McCormack JR. The management of mid-portion achilles tendinopathy with astym(R) and eccentric exercise: a case report. Int J Sports Phys Ther. 2012 Dec;7(6):672-7. PMID 23316430
- [Background] Henry P, Panwitz B, Wilson J. Rehabilitation of a Post-surgical Patella Fracture. Physiother. March 2000;86(3):139-142.
- [Background] McCrea EC, George SZ. Outcomes following augmented soft tissue mobilization for patients with knee pain: a case series. Orthop Phys Ther Pract. 2010;22(2):69-74.
- [Background] Haller KH, Helfst RH, Jr., Wilson JK, Sevier TL. Treatment of chronic elbow pain. Phys Ther Case Rep. 1999;2(5):195-200.
- [Background] Melham TJ, Sevier TL, Malnofski MJ, Wilson JK, Helfst RH Jr. Chronic ankle pain and fibrosis successfully treated with a new noninvasive augmented soft tissue mobilization technique (ASTM): a case report. Med Sci Sports Exerc. 1998 Jun;30(6):801-4. doi: 10.1097/00005768-199806000-00004. PMID 9624634
- [Background] Baker D, Wilson JK. Bilateral carpal tunnel syndrome in a piano teacher. Phys Ther Case Rep. 1999;2(2):73-76.
- [Background] Davidson CJ, Ganion LR, Gehlsen GM, Verhoestra B, Roepke JE, Sevier TL. Rat tendon morphologic and functional changes resulting from soft tissue mobilization. Med Sci Sports Exerc. 1997 Mar;29(3):313-9. doi: 10.1097/00005768-199703000-00005. PMID 9139169
- [Background] Gehlsen GM, Ganion LR, Helfst R. Fibroblast responses to variation in soft tissue mobilization pressure. Med Sci Sports Exerc. 1999 Apr;31(4):531-5. doi: 10.1097/00005768-199904000-00006. PMID 10211847
- [Background] Davies CC, Brockopp DY. Use of ASTYM® treatment on scar tissue following surgical treatment for breast cancer: a pilot study. Rehabil Oncology. 2010;28(3):3-12
- [Background] Sevier TL. ASTYM and the NFL. www.astym.com/Main 2011; http://blog.astym.com/blog/astym-3/astym-and-the-nfl. Accessed July 24th, 2012.
- [Background] Cook G. Athletic body in balance. Champaign, IL: Human Kinetics; 2003.
- [Background] Lockie RG, Schultz AB, Callaghan SJ, Jeffriess MD. The Relationship Between Dynamic Stability and Multidirectional Speed. J Strength Cond Res. 2016 Nov;30(11):3033-3043. doi: 10.1519/JSC.0b013e3182a744b6. PMID 23942170
- [Background] Health-Related Physical Fitness Testing and Interpretation In: Pescatello L, Riebe D, Thompson P, eds. American College of Sports Medicine's Guidelines for Exercise Testing and Prescription. Philadelphia, PA: Wolters Kluwer; 2014:60-109.
- [Background] General Principles of Exercise Prescription. In: Riche D, ed. American College of Sports Medicine's Guidelines for Exercise Testing and Prescription. Philadelphia, PA: Wolters Kluwer; 2014:164-166.
- [Background] Heyward VH, Gibson AL. Designing Cardiorespiratory Exercise Programs. Advanced Fitness Assessment and Exercise Prescription. Champaign, IL: Human Kinetics; 2014:131, 393-396.
- [Background] Heyward VH, Gibson AL. Assessing Cardiorespiratory Fitness. Advanced Fitness Assessment and Exercise Prescription. Champaign, IL: Human Kinetics; 2014:83-86.
- [Background] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777
- [Background] Buckthorpe M, Morris J, Folland JP. Validity of vertical jump measurement devices. J Sports Sci. 2012;30(1):63-9. doi: 10.1080/02640414.2011.624539. Epub 2011 Nov 23. PMID 22111944
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Sevier TL. What is IASTM? Is it different than Astym? www.astym.com/Main [Website]. 2013; http://blog.astym.com/blog/astym-3/what-is-iastm-is-it-different-than-astym. Accessed March 1st, 2013.
- [Background] Sevier TL. Astym and Soft Tissue Mobilization are Very Different. www.astym.com/Main [Website]. 2011; http://astym.com/blog/2011/06/27/astym-and-soft-tissue-mobilization-are-very-different.html#more-500006. Accessed September 26th, 2015.
- [Background] Sevier TL. Astym vs. IASTM: How Are They Different www.astym.com/Main 2010; http://astym.com/blog/2010/09/23/astym-vs-iastm-graston-sastm-etc-how-they-are-different.html#more-500117. Accessed September 26th, 2015.
- [Background] Cook G, Burton L, Kiesel K, Rose G, Bryant MF. Movement Functional Movement Systems: Screening, Assessment, and Corrective Strategies. Aptos, CA: On Target Publications; 2010.
- [Background] Potach D, Grindstaff T. Rehabilitation and Reconditioning. Essentials of Strength Training and Conditioning. 3rd ed: Human Kinetics; 2008.
- [Background] Steindler A. Kinesiology of the Human Body Under Normal and Pathological Conditions. Springfield; IL: C.C. Thomas; 1955.
- [Background] Prentice WE. Rehabilitation techniques in sports medicine and athletic training. 4th ed. Boston, MA: McGraw-Hill; 2004.
- [Background] Davies CC, Brockopp D, Moe K. Astym therapy improves function and range of motion following mastectomy. Breast Cancer (Dove Med Press). 2016 Mar 8;8:39-45. doi: 10.2147/BCTT.S102598. eCollection 2016. PMID 27022302
- [Background] What is The Stick? [Website]. 2014; http://thestick.com/info/about/. Accessed March 29, 2014
- [Background] The Stick Instructions. [The Stick Web Site]. http://www.thestick.co.nz/how-to-use.html. Accessed July 7, 2012.